CLINICAL TRIAL: NCT02650921
Title: A Randomized, Evaluator Blinded, Split-hand Study to Evaluate the Effectiveness and Safety of Restylane Lyft With Lidocaine Compared to no Treatment for Injection in the Dorsal Hand to Correct Volume Deficit
Brief Title: Effectiveness and Safety of Restylane Lyft With Lidocaine in the Dorsal Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43USH1501
Record Dates: First submitted 2015-12-21; First posted 2016-01-08 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2018-11

CONDITIONS: Volume Deficit in the Hand

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Restylane Lyft with Lidocaine (Experimental)
  Interventions: Device: Restylane Lyft with Lidocaine
- No Intervention (No Intervention)

INTERVENTIONS:
Device: Restylane Lyft with Lidocaine — An injectable gel of Hyaluronic Acid and Lidocaine
  Arms: Restylane Lyft with Lidocaine

SUMMARY:
This is a randomized, evaluator-blind, split hand, multi-center study of the effectiveness and safety or Restylane Lyft with Lidocaine compared to no treatment for injection in the dorsal hand to correct volume deficits.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects willing to comply with the requirements of the study and providing a signed written informed consent including release of copyright of hand images.
* Males or females, 22 years of age or older
* Willing and able to perform hand functionality tests .

Key Exclusion Criteria:

* History of allergy or hypersensitivity to injectable HA gel or to gram positive bacterial proteins.
* History of allergy or hypersensitivity to lidocaine or other amide type anesthetics.
* Previous hand surgery including sclerotherapy, or history of hand trauma.
* Advanced photo aged/ photo damaged skin or skin condition with very crinkled or fragile skin on the dorsal hands.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Vista, California
  - Boulder, Colorado
  - Englewood, Colorado
  - Boca Raton, Florida
  - St Louis, Missouri
  - Mount Kisco, New York
  - New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Moradi A, Allen S, Bank D, Marmur E, Fagien S, Glaser DA, Maguire C, Cohen JL. A Prospective, Multicenter, Randomized, Evaluator-Blinded, Split-Hand Study to Evaluate the Effectiveness and Safety of Large-Gel-Particle Hyaluronic Acid with Lidocaine for the Correction of Volume Deficits in the Dorsal Hand. Plast Reconstr Surg. 2019 Oct;144(4):586e-596e. doi: 10.1097/PRS.0000000000006070. PMID 31568288

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Hands
Groups:
- All Subjects: Subjects randomized to treatment with Restylane Lyft with Lidocaine in one hand and no treatment in the other
Period: Overall Study
Arm/Group | All Subjects
Started | 92; 184 Hands
Completed | 84; 168 Hands
Not Completed | 8; 16 Hands
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 1
Not completed — Due to Medical Condition | 1

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Restylane Lyft With Lidocaine: Restylane Lyft with Lidocaine: An injectable gel of Hyaluronic Acid and Lidocaine;
  Subjects were randomized to receive Restylane Lyft with Lidocaine in either the right or left hand.
Arm/Group | Restylane Lyft With Lidocaine
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 5
  White | 71
  More than one race | 5
  Unknown or Not Reported | 0
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  FST I (Always burns, never tans) | 4
  FST II (Usually burns, tans with difficulty) | 21
  FST III (Sometimes mild burns, gradually tans) | 39
  FST IV (Rarely burns, tans with ease) | 12
  FST V (Very rarely burns, tans with ease) | 7
  FST VI (Never burns, tans very easily) | 2
Hand Grading Scale - Treated hand [Count of Participants; unit: Participants] — Hand grading scale assessed by the Blinded evaluator
  Participants
    0 (No loss of fatty tissue) | 0
    1 (Mild loss of fatty tissue) | 0
    2 (Moderate loss of fatty tissue) | 27
    3 (Severe loss of fatty tissue) | 31
    4 (Very severe loss of fatty tissue) | 27
Hand Grading Scale - Fellow Hand [Count of Participants; unit: Participants] — Hand grading scale assessed by the Blinded evaluator
  Participants
    0 (No loss of fatty tissue) | 0
    1 (Mild loss of fatty tissue) | 0
    2 (Moderate loss of fatty tissue) | 18
    3 (Severe loss of fatty tissue) | 39
    4 (Very severe loss of fatty tissue) | 28

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate Using Validated Hand Grading Scale
Description: A responder is defined as a hand with at least one improvement from baseline.
Time Frame: 12 Weeks
Population: ITT population
Measure: Count of Participants; unit: Participants
Groups:
- Restylane Lyft With Lidocaine: Hands randomized to treatment with Restylane Lyft with Lidocaine
- No Intervention: Hands randomized to no treatment
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 85 | 85
Participants
  Responder | 73 | 18
  Non-Responder | 12 | 67
Statistical Analysis 1: Comparison: Restylane Lyft With Lidocaine vs No Intervention; Test type: Superiority; p < 0.0001, McNemar; Difference in Responder Rate = 64.7, 95% CI 2-sided [53.3 to 76.1]

2. Secondary Outcome: Responder Rate Using Validated Hand Grading Scale
Description: A responder is defined as a hand with at least one point improvement from baseline
Time Frame: 16 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 83 | 83
Participants
  Responder | 76 | 16
  Non-Responder | 7 | 67
Statistical Analysis 1: Comparison: Restylane Lyft With Lidocaine vs No Intervention; Test type: Superiority; p < 0.0001, McNemar; Difference in Responder Rate = 72.3, 95% CI 2-sided [61.9 to 82.7]

3. Secondary Outcome: Responder Rate Using Validated Hand Grading Scale
Description: A responder is defined as a hand with at least one point improvement from baseline
Time Frame: 20 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 82 | 82
Participants
  Responder | 68 | 21
  Non-Responder | 14 | 61
Statistical Analysis 1: Comparison: Restylane Lyft With Lidocaine vs No Intervention; Test type: Superiority; p < 0.0001, McNemar; Difference in Responder Rate = 57.3, 95% CI 2-sided [44.8 to 69.8]

4. Secondary Outcome: Responder Rate Using Validated Hand Grading Scale
Description: A responder is defined as a hand with at least one point improvement from baseline.
Time Frame: 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 83 | 83
Participants
  Responder | 63 | 25
  Non-Responder | 20 | 58
Statistical Analysis 1: Comparison: Restylane Lyft With Lidocaine vs No Intervention; Test type: Superiority; p < 0.0001, McNemar; Difference in Responder Rate = 45.8, 95% CI 2-sided [32.3 to 59.3]

5. Secondary Outcome: Improvement in Hand as Evaluated by IPR
Description: Independent Photographic Reviewer's assessment of improvement (Yes/No)
Time Frame: 12 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 84 | 84
Participants
  Yes | 74 | 16
  No | 10 | 68

6. Secondary Outcome: Improvement in Hand as Evaluated by IPR
Description: Independent Photographic Reviewer's assessment of improvement (Yes/No)
Time Frame: 16 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 83 | 83
Participants
  Yes | 71 | 17
  No | 12 | 66

7. Secondary Outcome: Improvement in Hand as Evaluated by IPR
Description: Independent Photographic Reviewer's assessment of improvement (Yes/No)
Time Frame: 20 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 82 | 82
Participants
  Yes | 57 | 13
  No | 25 | 69

8. Secondary Outcome: Improvement in Hand as Evaluated by IPR
Description: Independent Photographic Reviewer's assessment of improvement (Yes/No)
Time Frame: 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 83 | 83
Participants
  Yes | 71 | 18
  No | 12 | 65

9. Secondary Outcome: GAIS by Treating Investigator
Description: Global Aesthetic Improvement Scale
Time Frame: 12 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 84 | 84
Participants
  Very much improved | 40 | 0
  Much improved | 37 | 0
  Improved | 6 | 0
  No change | 1 | 84
  Worse | 0 | 0

10. Secondary Outcome: GAIS by Treating Investigator
Description: Global Aesthetic Improvement Scale
Time Frame: 16 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 83 | 83
Participants
  Very much improved | 40 | 0
  Much improved | 36 | 1
  Improved | 5 | 0
  No change | 1 | 82
  Worse | 1 | 0

11. Secondary Outcome: GAIS by Treating Investigator
Description: Global Aesthetic Improvement Scale
Time Frame: 20 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 82 | 82
Participants
  Very much improved | 33 | 0
  Much improved | 40 | 0
  Improved | 8 | 0
  No change | 1 | 82
  Worse | 0 | 0

12. Secondary Outcome: GAIS by Treating Investigator
Description: Global Aesthetic Improvement Scale
Time Frame: 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 83 | 83
Participants
  Very much improved | 24 | 1
  Much improved | 45 | 0
  Improved | 10 | 0
  No change | 3 | 82
  Worse | 1 | 0

13. Secondary Outcome: Evaluate GAIS by Subjects
Description: Global Aesthetic Improvement Scale
Time Frame: 12 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 84 | 84
Participants
  Very much improved | 34 | 0
  Much improved | 30 | 0
  Improved | 18 | 0
  No change | 1 | 84
  Worse | 1 | 0

14. Secondary Outcome: Evaluate GAIS by Subjects
Description: Global Aesthetic Improvement Scale
Time Frame: 16 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 83 | 83
Participants
  Very much improved | 27 | 0
  Much improved | 31 | 0
  Improved | 21 | 2
  No change | 4 | 81
  Worse | 0 | 0

15. Secondary Outcome: Evaluate GAIS by Subjects
Description: Global Aesthetic Improvement Scale
Time Frame: 20 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 82 | 82
Participants
  Very much improved | 21 | 0
  Much improved | 34 | 1
  Improved | 22 | 0
  No change | 5 | 80
  Worse | 0 | 1

16. Secondary Outcome: Evaluate GAIS by Subject
Description: Global Aesthetic Improvement Scale
Time Frame: 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine | No Intervention
Number analyzed (Participants) | 83 | 83
Participants
  Very much improved | 21 | 0
  Much improved | 26 | 1
  Improved | 30 | 1
  No change | 5 | 80
  Worse | 1 | 1

17. Secondary Outcome: Question 1 From Subject Satisfaction Questionnaire
Description: Question 1: I am happier with the overall appearance of my treated hand compared to my untreated hand
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Groups:
- Restylane Lyft With Lidocaine: Subjects that received treatment with Restylane Lyft with Lidocaine
Arm/Group | Restylane Lyft With Lidocaine
Number analyzed (Participants) | 84
Participants
  Agree | 77
  Do Not Agree | 7

18. Secondary Outcome: Question 2 From Subject Satisfaction Questionnaire
Description: Question 2: My treated hand appears more attractive than my untreated hand
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine
Number analyzed (Participants) | 84
Participants
  Agree | 74
  Do Not Agree | 10

19. Secondary Outcome: Question 3 From Subject Satisfaction Questionnaire
Description: Question 3: My treated hand looks more youthful than my untreated hand
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine
Number analyzed (Participants) | 84
Participants
  Agree | 75
  Do Not Agree | 9

20. Secondary Outcome: Question 4 From Subject Satisfaction Questionnaire
Description: Question 4: My treated hand feels softer than my untreated hand
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine
Number analyzed (Participants) | 84
Participants
  Agree | 44
  Do Not Agree | 40

21. Secondary Outcome: Question 5 From Subject Satisfaction Questionnaire
Description: Question 5: The skin on my treated hand appears tighter than on my untreated hand
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine
Number analyzed (Participants) | 84
Participants
  Agree | 64
  Do Not Agree | 20

22. Secondary Outcome: Question 6 From Subject Satisfaction Questionnaire
Description: Question 6: My treated hand looks less bony than my untreated hand
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine
Number analyzed (Participants) | 84
Participants
  Agree | 78
  Do Not Agree | 6

23. Secondary Outcome: Question 7 From Subject Satisfaction Questionnaire
Description: Question 7: The veins on my treated hand are less apparent compared to my untreated hand
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine
Number analyzed (Participants) | 84
Participants
  Agree | 81
  Do Not Agree | 3

24. Secondary Outcome: Question 8 From Subject Satisfaction Questionnaire
Description: Question 8: My treated hand appears at least 5 years younger than my untreated hand
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine
Number analyzed (Participants) | 84
Participants
  Agree | 59
  Do Not Agree | 25

25. Secondary Outcome: Question 9 From Subject Satisfaction Questionnaire
Description: Question 9: My treated hand appears at least 10 years younger than my untreated hand
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine
Number analyzed (Participants) | 84
Participants
  Agree | 26
  Do Not Agree | 58

26. Secondary Outcome: Question 10 From Subject Satisfaction Questionnaire
Description: Question 10: The skin on my treated hand appears hydrated
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine
Number analyzed (Participants) | 83
Participants
  Agree | 57
  Do Not Agree | 26

27. Secondary Outcome: Question 11 From Subject Satisfaction Questionnaire
Description: Question 11: The treatment result looks natural
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine
Number analyzed (Participants) | 84
Participants
  Agree | 80
  Do Not Agree | 4

28. Secondary Outcome: Question 12 From Subject Satisfaction Questionnaire
Description: Question 12: I would recommend this treatment to a friend
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine
Number analyzed (Participants) | 84
Participants
  Agree | 71
  Do Not Agree | 13

29. Secondary Outcome: Question 13 From Subject Satisfaction Questionnaire
Description: Question 13: I would have another treatment to maintain these results
Time Frame: Week 12
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Lyft With Lidocaine
Number analyzed (Participants) | 84
Participants
  Agree | 65
  Do Not Agree | 19

ADVERSE EVENTS:
Time Frame: 32 weeks
Description: AEs were collected by subject direct report, subject interview, or obtained from signs/symptoms detected during examination.
Arm/Group | Restylane Lyft With Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/89
Serious Adverse Events (participants affected / at risk) | 0/89
Other Adverse Events (participants affected / at risk) | 37/89
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Lyft With Lidocaine (N=89)
Peripheral Swelling (General disorders) | 4 (6)
Laceration (Injury, poisoning and procedural complications) | 6 (6)
Scratch (Injury, poisoning and procedural complications) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7)
Bronchitis (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Tooth Infection (Infections and infestations) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (3)
Thermal Burn (Injury, poisoning and procedural complications) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Vitreous Detachment (Eye disorders) | 1 (1)
Cyst Rupture (General disorders) | 1 (1)
Device Failure (General disorders) | 1 (1)
Facial Pain (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Chronic Sinusitis (Infections and infestations) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1)
Animal Scratch (Injury, poisoning and procedural complications) | 1 (1)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1)
Eye Injury (Injury, poisoning and procedural complications) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1)
Nail Injury (Injury, poisoning and procedural complications) | 1 (1)
Blood Cholesterol Increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No